CLINICAL TRIAL: NCT04289402
Title: Modulating Brain Activity to Improve Cognitive-motor Function in Alzheimer's Disease
Brief Title: Individualized Brain Stimulation to Improve Mobility in Alzheimer's Disease
Acronym: ISTIM-AD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Brad Manor, Assistant Scientist II; Director, Mobility and Brain Function Lab, Hinda and Arthur Marcus Institute for Aging Research, Hebrew SeniorLife
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3P30AG031679-09S1 (NIH)
Record Dates: First submitted 2020-02-13; First posted 2020-02-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Dementia; Presenile Alzheimer Dementia; Aging
Keywords: Aging
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a single site, sham-controlled, double-blinded, randomized trial of tDCS. Participants will complete baseline cognitive and physical functioning assessments, as well as a structural MRI of the brain. They will then be assigned to a two-week, 10-session intervention of either personalized tDCS sham (i.e., control) stimulation, via permuted block randomization stratified by sex to ensure that equal number of men and women are randomized to each intervention arm.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study personnel administering tDCS and the participants will not be aware of tDCS intervention arm assignment. The investigators will ensure double-blinding by programming the tDCS software with intervention-specific stimulation codes, as supplied by personnel uninvolved in data collection prior to study initiation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Personalized tDCS (Experimental): Baseline MRIs will enable personalization of tDCS via current flow modeling for optimization to each participant with the goal of generating an average electric field of 0.25 V/m within their identified left dlPFC. The direct current delivered by any one electrode will not exceed 2.0 mA and the total amount of current from all electrodes will not exceed 4 mA. Each 20-minutes session will begin and end with a 60-second ramp up/down of current amplitude to maximize comfort.
  Interventions: Other: Personalized tDCS
- Active-Sham (Sham Comparator): The investigators will use an active sham in which very low-level currents (0.5 mA total) will be transferred between electrodes in close proximity on the scalp throughout the entire 20-minute session. This intervention will be optimized to each participant to deliver currents designed to not significantly influence their cortical tissue, but still mimic the cutaneous sensations induced by tDCS.
  Interventions: Other: Active-Sham

INTERVENTIONS:
Other: Personalized tDCS — The participant will receive 10, 20-minutes sessions of personalized tDCS Monday-Friday, at approximately the same time of day, over two consecutive weeks.
  Arms: Personalized tDCS
Other: Active-Sham — The participant will receive 20, 20-minute sessions of active-sham stimulation Monday-Friday, at approximately the same time of day, over two consecutive weeks.
  Arms: Active-Sham

SUMMARY:
The objective of this study is to conduct a pilot, randomized sham-controlled trials to determine the feasibility and effects of a 10-session personalized tDCS intervention targeting the left dorsolateral prefrontal cortex on cognitive function, dual task standing and walking, and other metrics of mobility in 24 older adults with mild AD living in supportive housing.

DETAILED DESCRIPTION:
Beyond the profound impact on memory, Alzheimer's disease (AD) neuropathology, even in its early stages, affects the prefrontal lobes leading to executive dysfunction and mobility disturbances. Prefrontal cortex functions, including executive control, attention, and working memory, are known to decline with the progression of AD. In older adults, better performance on executive cognitive tasks is associated with greater activation of the left dorsolateral prefrontal cortex (dlPFC). Reduced activation within the dlPFC is believed to play a role in both the executive and physical functioning declines seen in AD, significantly contributing to loss of functional independence. In mild AD, an individual's state of executive functioning is a sensitive predictor of the ability to stand and walk safely, especially when performing additional cognitive tasks (i.e., dual tasking). Therefore, the investigators contend that by facilitating the excitability of the left dlPFC, some of the early cognitive and mobility impairments of AD may be reduced, ultimately leading to more functional independence, increased physical activity, and improved quality of life.

tDCS provides a noninvasive means of facilitating the excitability of the prefrontal cortex and its connected neural networks, and thus holds promise as a therapy to improve the executive control of cognition and mobility in older adults with mild AD. tDCS modulates cortical excitability by passing low-level currents through electrodes placed upon the scalp over the dlPFC. These currents induce electrical fields within the brain that in turn polarize neuronal populations and alter their likelihood of firing. The research team demonstrated in older adults aged 65 years and older with executive dysfunction and slow gait that 10 sessions of 20-minutes of tDCS targeting the left dlPFC improved cognitive and physical functioning for at least two weeks following the intervention. Considerable evidence, including our preliminary studies, now suggest that multi-session tDCS interventions targeting the dlPFC may induce measurable and meaningful improvements in cognitive and/or mobility outcomes in relatively healthy adults and in those with mild-to-moderate executive dysfunction. Still, the size and duration of tDCS-induced benefits in older adults with executive dysfunction have not been established. Moreover, to date, tDCS delivery has not attempted to account for interpersonal differences in older adults, particularly the high inter-individual variance in skin, skull, brain, and cerebrospinal fluid and how each of these characteristics impacts the current flow. Such personalization is now possible with the current flow modeling the investigators propose.

The overall aim of the study is to conduct a pilot, randomized sham-controlled trial to determine the feasibility and effects of a 10-session personalized tDCS intervention targeting the left dlPFC on cognitive function, dual task standing and walking, and other metrics of mobility in 24 older adults with mild AD living in supportive housing. The investigators will include personalized current flow modeling approach using baseline structural MRIs to determine the tDCS electrode placement and stimulation parameters to optimize current flow to each participant's brain. The investigators do not expect tDCS to revere the structural brain changes that result from AD, but instead maximize the function of remaining, intact brain neurons and frontal networks, and thereby improve functional outcomes in people suffering from the neurodegenerative process.

The investigators hypothesize that, in older adults 65 years and older with mild AD, a personalized tDCS intervention targeting the left dlPFC, as compared to sham, will mitigate dual task costs to the control of gait and standing posture and enhance executive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 65 and older living within supportive housing facilities
* Mild Alzheimer's disease (AD) defined by the combination of 1) at least mild cognitive impairment defined as a modified TICS score of ≤ 34, 2) informant-report of Instrumental Activities of Daily Living impairment as defined as a score of ≥ 6 on the NACC Functional Activities Questionnaire, and 3) a Clinical Dementia Rating score of 1.

Exclusion Criteria:

* Inability to secure informant participation
* Unwillingness to cooperate or participate in the study protocol
* An inability to ambulate without the assistance of another person (canes or walkers allowed)
* A clinical history of stroke, Parkinson's disease or parkinsonian symptoms, multiple sclerosis, normal pressure hydrocephalus, or other neurological conditions outside of mild AD.
* Any report of severe lower-extremity arthritis or physician-diagnosis of peripheral neuropathy
* Use of antipsychotics, anti-seizure, benzodiazepines, or other neuroactive medications
* Severe depression defined by a Center for Epidemiologic Studies Depression scale score greater than 16
* Any report of physician-diagnosis of schizophrenia, bipolar disorder, or other psychiatric illness
* Contraindications to MRI or tDCS, including reported seizure within the past two years, use of neuropsychological-active drugs, the risk of metal objects anywhere in the body, self-reported presence of specific implanted medical devices (e.g., deep brain stimulator, medication infusion pump, cochlear implant, pacemakers, etc.), or the presence of any active dermatological condition, such as eczema, on the scalp

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment efficiency | 1 year
  The number of residents that need to be screened in order to enroll one participant into the trial.
Retention | 1 year
  The percentage of enrolled participants who complete the trial.
Blinding | Immediately after intervention
  A blinding efficacy questionnaire will be used to record participant guesses of their assigned intervention (real or placebo), as well as the confidence of these guesses on a scale from 1=Not confident to 10=Extremely confident.
Montreal Cognitive Assessment (MoCA) total score | Change from baseline to two-week follow-up
  This common test assesses global cognitive function. Maximum score on the MoCA is 30 points (minimum = 0), with higher scores associated with better outcomes.
Dual task gait speed | Change from baseline to two-week follow-up
  This metric assesses the ability to control gait while performing a secondary cognitive task.
Dual task standing postural sway area | Change from baseline to two-week follow-up
  This metric assesses the ability to control standing posture while performing a secondary cognitive task.

SECONDARY OUTCOMES:
Trail making test A-B | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses cognitive executive function.
Digit Span | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This common test assesses working memory.
Digit Symbol Substitution Test | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This common test assesses sustained attention and motor speed.
Category and Phonemic Fluency Test | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This common test assesses word retrieval.
Hopkins Verbal Learning Test | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This common test assesses memory.
Dual task stride time variability | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses the ability to control gait while performing a secondary cognitive task.
Dual task standing postural sway speed | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses the ability to control standing posture while performing a secondary cognitive task.
Timed Up-and-Go | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses mobility.
Five-day accelerometry-based physical activity | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses the quantity and quality of habitual physical activity.
Centers for Epidemiologic Studies Depression Scale | Baseline, within 3 days after completion of the intervention, two weeks after completing the intervention
  This metric assesses mood.

CONTACTS AND LOCATIONS:
Overall Officials: Brad Manor, PhD, Principal Investigator — Hebrew SeniorLife
Locations (1):
- Hebrew Rehabilitation Center, Roslindale, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The HSL Institute for Aging Research will promote the development of new research and new investigators by making the data available to outside investigators. The database will include longitudinal demographic, clinical, functional, physiologic, and brain imaging data, from all participants.
  All data will be stripped of primary identifiers and entered into a master database. All data collection procedures, variable definitions and codes, field locations, and frequencies will be documented in a separate file.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The investigators will make the data and associated documentation available once summary data are published or otherwise made available, starting six months after publication.
Access Criteria: The investigators will make the data and associated documentation available to users only under a data-sharing agreement that provides for: 1) a commitment to using data only for research purposes and not to identify any particular participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed. The availability of data will be advertised over the Internet through websites maintained by Hebrew SeniorLife and Harvard Medical School.
  All investigators wishing to access the data will submit a brief proposal describing their research project, data needs, regulatory approvals, and mechanisms to assure patient confidentiality. Upon affirmative review by the Principal Investigator and co-investigators of this study, a data-sharing agreement will be signed and the requesting investigators will be given a working data file and appropriate documentation.